CLINICAL TRIAL: NCT07189650
Title: Collection of Quantitative Data on Liver Fat Content Obtained From Ultrasound Attenuation (QAI) and Scattering (QSI) Imaging and From Liver Fat Fraction Values Obtained by Magnetic Resonance Imaging With Proton Density Technique (MRI-PDFF)
Brief Title: Pilot Study for Collecting Data on Liver Adipose Content in Adults by Ultrasound Attenuation and Scattering Imaging and MRI Proton-density
Acronym: QAI_QSI_MRI
Status: Not yet recruiting | Type: Observational
Sponsor: Esaote S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP000004
Record Dates: First submitted 2025-09-12; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Dysfunction-Associated Liver Disease
Keywords: Metabolic Dysfunction-Associated Liver Disease,; MASLD; Ultrasound - Tissue attenuation Imaging; Ultrasound - Tissue scatter imaging; MRI - Proton Density Fat Fraction; QAI; QSI; MRI-PDFF

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single Cohort: not vulnerable, adult subjetcs affected by MASLD (Metabolic Dysfunction-Associated Liver Disease)
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Proton Density Fat Fraction Magnetic Resonance Imaging (MRI-PDFF )

SUMMARY:
The aim of this single-center, prospective, pilot study is to acquire data on liver adipose content in a population of adult patients affected by MASLD (Metabolic Dysfunction-Associated Liver Disease).

Ultrasound attenuation (QAI) and scattering (QSI) imaging parameters will be acquired.

Fat percentage parameters, obtained from magnetic resonance imaging with proton density technique (MRI-PDFF), will be acquired as well and they will be considered as reference method and gold standard.

The study is initiated for exploratory and research purposes. The study will enroll 30 consecutive, non-vulnerable adult participants who are scheduled to undergo upper abdominal ultrasound (Intervention A) as part of their standard clinical evaluation for the diagnosis and/or management of steatotic liver disease (SLD).

Eligible participants will be invited to provide informed consent to undergo an additional, non-invasive imaging procedure (Intervention B), consisting of magnetic resonance imaging with proton density fat fraction (MRI-PDFF) quantification

DETAILED DESCRIPTION:
The primary endpoint of this exploratory study is to acquire data on liver adipose content in a population of adult patients affected by MASLD for comparing Ultrasound Imaging (QAI and QSI) and MRI (MRI-PDFF) methods

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis or suspected steatosic liver disease. The diagnosis may be suspected in the presence of concomitant conditions, such as (but not limited to) obesity, type 2 diabetes, pro-atherogenic dyslipidemia (hypertriglyceridemia, low HDL cholesterol), and metabolic syndrome;
* Patients for whom an upper abdominal ultrasound is indicated as part of the clinical workup for the diagnosis and/or treatment of steatosic liver disease.

Exclusion Criteria:

* Contraindications to MRI (patients with a pacemaker, metal implants, pregnant patients, claustrophobia, physical inability to perform the exam due to constitution);
* Inappropriate alcohol consumption (>30 g/day for men and >20 g/day for women);
* Viral liver disease (HBV, HCV, HIV);
* Other forms of metabolic/autoimmune/cholestatic or storage liver disease e.g., primary biliary cholangitis, sclerosing cholangitis, hemochromatosis, Wilson's disease);
* History of hepatocellular carcinoma or other forms of malignancy;
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients affected by MASLD (Metabolic Dysfunction-Associated Liver Disease)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Exploratory comparison of Ultrasound Imaging findings (Tissue Attenuation Imaging and Tissue Scatter Imaging) with MRI one (MRI-PDFF, considered as reference) in evaluating liver adipose content | through study completion, an average of 1 year
  Exploratory and preliminary comparison of the findings obtained assessing liver adipose content in a population of adult patients affected by MASLD (Metabolic Dysfunction-Associated Liver Disease) utilizing Ultrasound Imaging (Tissue Attenuation Imaging and Tissue Scatter Imaging) technologies and MRI one (MRI-PDFF). The latter is considered as reference technology and gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Garcovich, MD, PhD, Principal Investigator — UOSD Ecografia Diagnostica e Interventistica - Fondazione Policlinico Universitario Gemelli IRCCS, Rome (Italy)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers as this is a pilot-exploratory study that seek to generate hypotheses rather than a confirmatory study testing a specific, predetermined hypothesis with the goal of providing conclusive evidence in support of it.

REFERENCES:
- [Background] Han A, Andre MP, Deiranieh L, Housman E, Erdman JW Jr, Loomba R, Sirlin CB, O'Brien WD Jr. Repeatability and Reproducibility of the Ultrasonic Attenuation Coefficient and Backscatter Coefficient Measured in the Right Lobe of the Liver in Adults With Known or Suspected Nonalcoholic Fatty Liver Disease. J Ultrasound Med. 2018 Aug;37(8):1913-1927. doi: 10.1002/jum.14537. Epub 2018 Jan 23. PMID 29359454
- [Background] Noureddin M, Lam J, Peterson MR, Middleton M, Hamilton G, Le TA, Bettencourt R, Changchien C, Brenner DA, Sirlin C, Loomba R. Utility of magnetic resonance imaging versus histology for quantifying changes in liver fat in nonalcoholic fatty liver disease trials. Hepatology. 2013 Dec;58(6):1930-40. doi: 10.1002/hep.26455. Epub 2013 Oct 17. PMID 23696515
- [Background] Ferraioli G, Berzigotti A, Barr RG, Choi BI, Cui XW, Dong Y, Gilja OH, Lee JY, Lee DH, Moriyasu F, Piscaglia F, Sugimoto K, Wong GL, Wong VW, Dietrich CF. Quantification of Liver Fat Content with Ultrasound: A WFUMB Position Paper. Ultrasound Med Biol. 2021 Oct;47(10):2803-2820. doi: 10.1016/j.ultrasmedbio.2021.06.002. Epub 2021 Jul 18. PMID 34284932
- [Background] Rockey DC, Caldwell SH, Goodman ZD, Nelson RC, Smith AD; American Association for the Study of Liver Diseases. Liver biopsy. Hepatology. 2009 Mar;49(3):1017-44. doi: 10.1002/hep.22742. No abstract available. PMID 19243014
- [Background] Cholongitas E, Senzolo M, Standish R, Marelli L, Quaglia A, Patch D, Dhillon AP, Burroughs AK. A systematic review of the quality of liver biopsy specimens. Am J Clin Pathol. 2006 May;125(5):710-21. doi: 10.1309/W3XC-NT4H-KFBN-2G0B. PMID 16707372
- [Background] Dasarathy S, Dasarathy J, Khiyami A, Joseph R, Lopez R, McCullough AJ. Validity of real time ultrasound in the diagnosis of hepatic steatosis: a prospective study. J Hepatol. 2009 Dec;51(6):1061-7. doi: 10.1016/j.jhep.2009.09.001. Epub 2009 Sep 20. PMID 19846234
- [Background] Tamaki N, Ajmera V, Loomba R. Non-invasive methods for imaging hepatic steatosis and their clinical importance in NAFLD. Nat Rev Endocrinol. 2022 Jan;18(1):55-66. doi: 10.1038/s41574-021-00584-0. Epub 2021 Nov 23. PMID 34815553
- [Background] Eslam M, Sanyal AJ, George J. Toward More Accurate Nomenclature for Fatty Liver Diseases. Gastroenterology. 2019 Sep;157(3):590-593. doi: 10.1053/j.gastro.2019.05.064. Epub 2019 May 31. No abstract available. PMID 31158374
- [Background] Loomba R, Sanyal AJ. The global NAFLD epidemic. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):686-90. doi: 10.1038/nrgastro.2013.171. Epub 2013 Sep 17. PMID 24042449
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. J Hepatol. 2016 Jun;64(6):1388-402. doi: 10.1016/j.jhep.2015.11.004. Epub 2016 Apr 7. No abstract available. PMID 27062661
- [Background] Ress C, Kaser S. Mechanisms of intrahepatic triglyceride accumulation. World J Gastroenterol. 2016 Jan 28;22(4):1664-73. doi: 10.3748/wjg.v22.i4.1664. PMID 26819531
- [Background] Younossi ZM, Blissett D, Blissett R, Henry L, Stepanova M, Younossi Y, Racila A, Hunt S, Beckerman R. The economic and clinical burden of nonalcoholic fatty liver disease in the United States and Europe. Hepatology. 2016 Nov;64(5):1577-1586. doi: 10.1002/hep.28785. Epub 2016 Sep 26. PMID 27543837
- [Background] Browning JD, Szczepaniak LS, Dobbins R, Nuremberg P, Horton JD, Cohen JC, Grundy SM, Hobbs HH. Prevalence of hepatic steatosis in an urban population in the United States: impact of ethnicity. Hepatology. 2004 Dec;40(6):1387-95. doi: 10.1002/hep.20466. PMID 15565570